CLINICAL TRIAL: NCT04495374
Title: Use of Oral Pregabalin as Preemptive Analgesia in Abdominal Hysterectomy: Evaluation of Postoperative Pain and Opioid Consumption
Brief Title: Oral Pregabalin as Preemptive Analgesia in Abdominal Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to an atypical health scenario caused by the COVID-19 pandemic
Sponsor: Universidade Federal de Alfenas (Other)
Responsible Party: Principal Investigator, Larissa Helena Lobo Torres Pacheco, Principal Investigator, Universidade Federal de Alfenas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3.334.050
Record Dates: First submitted 2020-07-24; First posted 2020-07-31 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative; Analgesia; Gabapentin Adverse Reaction; Opioid Abuse
Keywords: postoperative pain; multimodal analgesia; pregabalin; preemptive analgesia; abdominal hysterectomy; gabapentins
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Opioid-Related Disorders | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P(0) - Placebo (Placebo Comparator): Patients were randomly allocated to Group P(0) - Placebo by a double blind randomized study. Group P(0) received two placebo tablets as medication, 02h before the start of the anesthesic-surgical procedure in identical sealed envelops, only identified as medication A or B
  Interventions: Other: Placebo
- Group P(1) - Pregabalin 300mg (Experimental): Patients were randomly allocated to Group P(1) - Pregabalin 300mg by a double blind randomized study. Group P(1) received two tablets of pregabalin 150mg, 02h before the start of the anesthesic-surgical procedure in identical sealed envelops, only identified as medication A or B
  Interventions: Drug: Pregabalin 300mg

INTERVENTIONS:
Drug: Pregabalin 300mg — Group P1 will receive a 300 mg tablet of pregabalin, 02h before the surgical procedure
  Other Names: Preemptive analgesia
  Arms: Group P(1) - Pregabalin 300mg
Other: Placebo — Group P0 will receive a placebo tablet, 02h before the surgical procedure
  Other Names: Controls
  Arms: Group P(0) - Placebo

SUMMARY:
Postoperative pain affects 80% of surgical patients and is one of the main negative symptoms resulting from surgery. It impairs the recovery of patient since it is related to chronic pain, nausea and vomiting and longer hospital stay, generating higher cost to the health system. Thus, the use of new methods to control postoperative pain is recommended and multimodal analgesia, an opioid-sparing strategies, has been widely used by several researchers. Studies show that gabapentins have beneficial effects on postoperative pain control when used as pre-anesthetic medication, also showing a reduction in opioid consumption, with few adverse effects. Among gynecological surgeries, abdominal hysterectomy is one of the procedures that generates the highest degree of acute postoperative pain. Thus, the aim of the present study is to investigate the effect of oral pregabalin (300 mg) two hours before abdominal hysterectomy procedures on postoperative pain. This study is a randomized, double-blind, placebo controlled clinical trial. Patients submitted to abdominal hysterectomy for benign pathologies will be selected and divided into two groups: the placebo controlled group (P0) and the pregabalin 300 mg group (P1). Group P0 will receive a placebo tablet one hour before the procedure, while group P1 will receive a 300 mg tablet of pregabalin identical to the placebo tablet. The reduction of postoperative pain and the best quality of patient recovery will be evaluated using the Visual Analogue Pain Scale (VAS) and the McGill Pain Questionnaire. Also, it will be evaluated the consumption of opioids as a rescue analgesic medication and the presence of adverse effects such as nausea and vomiting.

DETAILED DESCRIPTION:
The sample population of this study is 102 female patients (50 already included in the study), who have undergone abdominal hysterectomy surgery for benign conditions, with or without joint oophorectomy / salpingectomy. The patients received spinal anesthesia, at hospital "Santa Casa de Alfenas" - Minas Gerais / Brazil ("Casa de Caridade Nossa Senhora do Perpétuo Socorro"). All surgeries were performed by the same team of surgeons.

All patients were evaluated and followed from the preoperative period, up to 24 hours postoperatively, passing through the intraoperative period. During all stages, patients were assisted by a properly trained multi-professional team, consisting of a doctor, nurse and nursing technician.

For the patient to be included in the study, she must have understood and agreed with the informed consent form that was explained in detail to all possible candidates in the preoperative period.

This is a double blind randomized study. The patients were randomly allocated to 02 groups, in which Group 1 received medication A (designated in the study as medication 1), whereas Group 2 received medication B (designated in the study as medication 2).

Study participants and researchers were blinded as to the use of drug / placebo to avoid measurement bias. To carry out the blinding process, an external researcher was assigned to randomize the groups and prepare the pills in opaque and closed envelopes characterized only by a control identification (A or B), which is known only to this researcher. Patients in both groups received identical sealed envelopes, 02h before the start of the anesthetic procedure, only identified as medication A or B, which contained two pills in each envelope. A second researcher is responsible for collecting data and monitoring the patient from the intraoperative period up to 24 hours after discharge from the post-anesthetic recovery room (PARR).

In the operating room, venoclysis was performed with jelco No. 18 or No. 20, and an infusion of 08 ml.kg-1 of crystalloid solution (lactated ringer). The patients were properly monitored with pulse oximetry, cardioscope, and non-invasive blood pressure monitor. After monitoring, patients were premedicated with intravenous (IV) midazolam at a dosage of 0.03 mg.kg1.

To perform spinal anesthesia, the patients were seated on the surgical stretcher by the nursing team. Asepsis and antisepsis were performed at the puncture site with alcoholic chlorhexidine solution. After placement of sterile drapes, local anesthesia was performed with 2.0% lidocaine without vasoconstrictor. The first attempt at subarachnoid puncture was performed, using the median technique, between the intervertebral levels L3-L4 or L4-L5 or L5-S1, with a 25 gauge Quincke needle for subarachnoid anesthesia. If there was a technical difficulty in the puncture, the paramedian puncture technique was chosen. The confirmation of the correct puncture was based on the aspiration of cerebrospinal fluid. Anesthesia was performed with the local anesthetic 0.5% bupivacaine at a dosage of 0.3 mg.kg-1, injected from a 5 ml disposable syringe. After anesthesia, the patients were placed in the supine position, and the correct level of anesthesia was proven with thermal sensitivity tests using cotton soaked with alcoholic solution. After the anesthesia reached the sensory level of the T4 thoracic vertebra, the surgical team was allowed to start the procedure. Prior to the beginning of the surgical incision, a delayed bladder probe was performed in all patients according to the surgeon's indication.

Hemodynamic changes in blood pressure were controlled with the use of vasoactive medications such as ephedrine or metaraminol. For prophylaxis of postoperative nausea and vomiting (PONV) ondansetron was administered at a dosage of 4 mg intravenously (IV) 30 minutes before the end of surgery. Tenoxicam was prescribed for all patients at a dosage of 20 mg IV at regular intervals every 12 hours for the purpose of anti-inflammatory and analgesic action. For analgesic relief, dipyrone IV was also prescribed at a dosage of 50 mg.kg-1 at regular intervals every 6 hours. During the surgery, and also at the end of the surgery, the patients were evaluated for the degree of sedation using the Ramsay sedation scale as a basis.

At the end of the surgery, the patients were referred to the post-anaesthesia care unit, where they were monitored again, and went through the pain assessment process using the visual analog scale (VAS) in relation to pain at rest and "movement" (the patient was asked to perform the forced cough movement), through a direct question with scale demonstration. Pains characterized as mild (0 - 2 VAS) received no medication other than those already prescribed; pain characterized as moderate (3 - 7 EVA) received IV morphine at a dosage of 0.025 mg.kg-1; and severe pain (8 - 10 VAS) received IV morphine at a dose of 0.05 mg.kg-1 every 01 h until analgesic control.

To consider themselves able to be discharged from the post-anaesthesia care unit for clinical follow-up in wards, patients should reach a score ≥ 9 on the modified Aldrete Scale and have VAS pain scores ≤ 2.

In the infirmary, patients were tested at regular intervals for pain intensity, by of a team of nurses trained and qualified to do so. The patients had pain classified as moderate (VAS ≥ 2 <8) or severe (VAS ≥ 8), receiving drugs with morphine IV in the dose of 1 mg and 2 mg respectively, according to the medical prescription.

24 h after discharge from the post-anaesthesia care unit, in the ward, all the patient was assessed by the same examiner who performed an assessment at the post-anaesthesia care unit, who stratified the patient again from the EVA and assessed using the McGill questionnaire.

During the entire hospitalization period, the use of central nervous system (CNS) depressant drugs (example: ketamine, droperidol, promethazine) and / or analgesic drugs that do not contain any study protocol was avoided. If some patients were medicated with these drugs, they were excluded from the study.

The data related to surgery (pre, trans and postoperative) were collected for statistical analysis, according to Annex II, in which a total duration of surgery in minutes; the total intravenous medication infused; the values of mean arterial pressure and heart rate in the pre, intra and postoperative period; a presence or not, as well as a quantity, of PONV in the post-anaesthesia care unit and after 24h; presence or not of dizziness as a possible side effect; among others.

All data selected through the study will be digitized and analyzed using the Statistic® 7.0 software. The data will be compared using repeated measures ANOVA, followed by Newman-Keuls post-hoc, being considered for p <0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will undergo elective abdominal hysterectomy surgery due to benign pathologies;
2. Be classified as physical status by the Society of Anesthesiologists (ASA) as ASA I (healthy individual) or ASA II (patient with mild and controlled systemic disease);

Exclusion Criteria:

1. Allergy or intolerance previously known to pregabalin or opioids;
2. Patients with chronic pain or fibromyalgia;
3. Patients on chronic opioid use;
4. Carriers of malignant neoplasms;
5. Pregnant women;
6. People with active uncontrolled cardiovascular disease;
7. Patients with kidney and / or liver disease;
8. Patients who have spinal deformities that make spinal anesthesia impossible;
9. Presence of coagulation disorders or anticoagulant therapy that cannot be suspended for surgery;
10. Presence of active sepsis.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 58 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa H Torres, PhD, Principal Investigator — Universidade Federal de Alfenas; Fabrício G Silva, BSc, Study Chair — Santa Casa de Alfenas; Carlos M de Barros, BSc, Study Chair — Universidade Federal de Alfenas; Marcia H Podestá, PhD, Study Chair — Universidade Federal de Alfenas; Carla S Ceron, PhD, Study Chair — Universidade Federal de Alfenas; Thayná C Silva, BSc, Study Chair — Santa Casa de Alfenas; Denismar A Nogueira, PhD, Study Chair — Universidade Federal de Alfenas; Tiago M Reis, PhD, Study Chair — Universidade Federal de Alfenas; Milena C Espósito, PhD, Study Chair — Universidade Federal de Alfenas; Danielle A Oliveira, BSc, Study Chair — Universidade Federal de Alfenas
Locations (1):
- Universidade Federal de Alfenas, Alfenas, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu J, Huang D, Li M, Wu C, Zhang J. Effects of a single dose of preoperative pregabalin and gabapentin for acute postoperative pain: a network meta-analysis of randomized controlled trials. J Pain Res. 2018 Nov 2;11:2633-2643. doi: 10.2147/JPR.S170810. eCollection 2018. PMID 30519075
- [Background] As-Sanie S, Till SR, Mowers EL, Lim CS, Skinner BD, Fritsch L, Tsodikov A, Dalton VK, Clauw DJ, Brummett CM. Opioid Prescribing Patterns, Patient Use, and Postoperative Pain After Hysterectomy for Benign Indications. Obstet Gynecol. 2017 Dec;130(6):1261-1268. doi: 10.1097/AOG.0000000000002344. PMID 29112660
- [Background] Farzi F, Naderi Nabi B, Mirmansouri A, Fakoor F, Atrkar Roshan Z, Biazar G, Zarei T. Postoperative Pain After Abdominal Hysterectomy: A Randomized, Double-Blind, Controlled Trial Comparing the Effects of Tramadol and Gabapentin as Premedication. Anesth Pain Med. 2016 Jan 17;6(1):e32360. doi: 10.5812/aapm.32360. eCollection 2016 Feb. PMID 27110531
- [Background] Ghai A, Gupta M, Hooda S, Singla D, Wadhera R. A randomized controlled trial to compare pregabalin with gabapentin for postoperative pain in abdominal hysterectomy. Saudi J Anaesth. 2011 Jul;5(3):252-7. doi: 10.4103/1658-354X.84097. PMID 21957402
- [Background] Kohli M, Murali T, Gupta R, Khan P, Bogra J. Optimization of subarachanoid block by oral pregabalin for hysterectomy. J Anaesthesiol Clin Pharmacol. 2011 Jan;27(1):101-5. PMID 21804717
- [Background] Main CJ. Pain assessment in context: a state of the science review of the McGill pain questionnaire 40 years on. Pain. 2016 Jul;157(7):1387-1399. doi: 10.1097/j.pain.0000000000000457. PMID 26713423
- [Background] Steinberg AC, Schimpf MO, White AB, Mathews C, Ellington DR, Jeppson P, Crisp C, Aschkenazi SO, Mamik MM, Balk EM, Murphy M. Preemptive analgesia for postoperative hysterectomy pain control: systematic review and clinical practice guidelines. Am J Obstet Gynecol. 2017 Sep;217(3):303-313.e6. doi: 10.1016/j.ajog.2017.03.013. Epub 2017 Mar 27. PMID 28351670
- [Background] Tulandi T, Krishnamurthy S, Mansour F, Suarthana E, Al-Malki G, Ballesteros LER, Moore A. A Triple-Blind Randomized Trial of Preemptive Use of Gabapentin Before Laparoscopic Hysterectomy for Benign Gynaecologic Conditions. J Obstet Gynaecol Can. 2019 Sep;41(9):1282-1288. doi: 10.1016/j.jogc.2018.11.019. Epub 2019 Jan 25. PMID 30686609
- [Background] Verret M, Lauzier F, Zarychanski R, Savard X, Cossi MJ, Pinard AM, Leblanc G, Turgeon AF. Perioperative use of gabapentinoids for the management of postoperative acute pain: protocol of a systematic review and meta-analysis. Syst Rev. 2019 Jan 16;8(1):24. doi: 10.1186/s13643-018-0906-3. PMID 30651123
- [Background] Yucel A, Ozturk E, Aydogan MS, Durmus M, Colak C, Ersoy MO. Effects of 2 different doses of pregabalin on morphine consumption and pain after abdominal hysterectomy: a randomized, double-blind clinical trial. Curr Ther Res Clin Exp. 2011 Aug;72(4):173-83. doi: 10.1016/j.curtheres.2011.06.004. PMID 24648587

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Started | 30 | 28
Completed | 28 | 27
Not Completed | 2 | 1
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Median (Standard Deviation); unit: years] | 41.5 (7.86) | 45 (4.15) | 43 (6.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 14 | 13 | 27
  Ethnicity: Black | 5 | 5 | 10
  Ethnicity: Brown | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain in Rest Assessed 24 Hours After Abdominal Hysterectomy Surgery Using the Visual Analog Scale (VAS)
Description: Postoperative pain assessment, 24 hours after abdominal hysterectomy surgery, in patients who used a single dose of pregabalin 300mg or placebo as preemptive analgesia, using the visual analog scale (VAS) consisting of a 10 cm (cm) line ) graduated in natural number intervals, starting at 0 (zero) until reaching 10 (ten), associated with the numbers, drawings related to the pain presented by the patient at the moment, in which the absence of pain (0 ) there is a happy face, and as the numerical value increases, the drawn face will represent the intensity of pain, up to the value of 10, where a face with crying characteristics is found, indicating greater pain.
Time Frame: End of the first postoperative day of abdominal hysterectomy surgery (24 hours after the end of surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Number analyzed (Participants) | 28 | 27
score on a scale | 5 (1.34) | 2 (1.19)

2. Primary Outcome: Postoperative Pain Assessed 24 Hours After Abdominal Hysterectomy Surgery, Using the McGill Pain Questionnaire
Description: Postoperative pain assessment, 24 hours after abdominal hysterectomy surgery, in patients who used a single 300mg dose of pregabalin or placebo as preemptive analgesia, using the McGill pain questionnaire, which consists of 20 word groups , and each group can contain from 2 to 6 descriptive words, these descriptors are placed in an increasing order of magnitude in relation to the intensity. The left of each word has a numerical value in an attempt to represent the intensity of the descriptor. For the analysis of the answers, the total number of words chosen in each subgroup by the patient was used to qualify his pain, the minimum value being equal to 0 (zero), if the patient chose not to choose any descriptor, and the maximum value would be 20, as the patient can choose only one descriptor for each subgroup. The quantitative pain index was also evaluated, which represents the sum of the values of each descriptor chosen by the patient, with a minimum value of 0 and a maximum of 78.
Time Frame: End of the first postoperative day of abdominal hysterectomy surgery (24 hours after the end of surgery)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Number analyzed (Participants) | 28 | 27
score on a scale | 28.5 (11) | 12 (10)

3. Primary Outcome: Postoperative Pain in Active Movement Assessed 24 Hours After Abdominal Hysterectomy Surgery Using the Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: End of the first postoperative day of abdominal hysterectomy surgery (24 hours after the end of surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Number analyzed (Participants) | 28 | 27
score on a scale | 7 (1.41) | 4 (1.39)

4. Secondary Outcome: Number of Doses of Opioids Used as Analgesic Rescue in the Postoperative Period
Description: Evaluation of the number of intravenous opioid doses used within 24 hours of postoperative abdominal hysterectomy surgery in patients who used pregabalin 300mg or not as preemptive analgesia
Time Frame: End of the first postoperative day of abdominal hysterectomy surgery (24 hours after the end of surgery)
Measure: Median (Standard Deviation); unit: number of doses
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Number analyzed (Participants) | 28 | 27
number of doses | 4 (1.91) | 2 (1.27)

5. Secondary Outcome: Time Required for the Use of the First Dose of Opioid as an Analgesic Rescue in the Postoperative Period
Description: • Evaluation of the time between the end of abdominal hysterectomy surgery and the patient's request for the use of the first dose of intravenous opioid as an analgesic rescue, comparing between patients who used or not pregabalin 300mg as preemptive analgesia
Time Frame: End of the first postoperative day of abdominal hysterectomy surgery (24 hours after the end of surgery)
Measure: Median (Standard Deviation); unit: Time in minutes
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Number analyzed (Participants) | 28 | 27
Time in minutes | 170 (177.6) | 106 (64.8)

6. Secondary Outcome: Number of Participants With Dizziness Between the Intervention and Control Groups
Description: • Assess the presence of adverse effects such as nausea and vomiting, itching and dizziness, comparing the intervention group that used pregabalin with the placebo group
Time Frame: End of the first postoperative day of abdominal hysterectomy surgery (24 hours after the end of surgery) and also immediately in the post-anesthetic recovery room
Measure: Count of Participants; unit: Participants
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
Number analyzed (Participants) | 28 | 27
Participants | 7 | 16

ADVERSE EVENTS:
Time Frame: Data related to adverse events were collected during the follow-up of patients from the preoperative period up to 24h postoperatively.
Description: Adverse events such as nausea and vomiting, pruritus, dizziness were evaluated during the entire follow-up of patients
Arm/Group | Group P(0) - Placebo | Group P(1) - Pregabalin 300mg
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 19/28 | 16/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group P(0) - Placebo (N=28) | Group P(1) - Pregabalin 300mg (N=27)
Dizziness (Nervous system disorders) | 7 | 16 — Dizziness is an adverse event that can commonly occur with the use of pregabalin
Nausea and vomiting (Gastrointestinal disorders) | 19 | 16 — The presence of nausea and vomiting is a common side effect of abdominal surgery, and its incidence may be increased by the use of opioids.
Pruritus (General disorders) | 1 | 2 — The presence of pruritus is a common adverse event in the use of opioids

LIMITATIONS AND CAVEATS:
Failure to monitor patients 24 hours after surgery to assess parameters such as chronic pain and home opioid consumption. All patients admitted to the study underwent abdominal hysterectomy, a surgery known to have higher pain rates, which makes it impossible for the results found to be used as a basis for patients undergoing laparoscopic hysterectomy or other types of surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT04495374/Prot_SAP_000.pdf